CLINICAL TRIAL: NCT02390726
Title: Fecal Microbiota Transplant in the Treatment of Ulcerative Colitis
Acronym: FMTUC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Peter L. Moses, MD, MD, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15373
Record Dates: First submitted 2015-02-19; First posted 2015-03-17 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Ulcerative Colitis, Active Moderate
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Sham Comparator): Sham FMT and Sham Microbial Maintenance plus standard therapy
  Interventions: Biological: Placebo
- Treatment (Experimental): FMT and microbial maintenance plus standard therapy
  Interventions: Biological: Fecal Microbiota Transplant

INTERVENTIONS:
Biological: Fecal Microbiota Transplant
  Arms: Treatment
Biological: Placebo
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Fecal Microbiota Transplant (FMT) for treating patients with mild to moderate Ulcerative Colitis (UC). Even with the expanding choices of medication for UC, physicians and patients are still in search of highly effective and safe medications with minimal side effects. FMT has been approved for the treatment of a bacterial infection called Clostridium difficile. In this setting, FMT has been proven to be an effective and safe alternative therapy with zero reported serious adverse events from patients that have had this treatment.

The providers that are conducting this study hypothesize that delivering microbes from a healthy human gut can help treat the damages caused by UC. This is done by "transplanting" fecal material, which contains a highly complex and dense community of healthy microbes, including bacteria, fungi and viruses. This collection of microbes is referred to as a microbiome. Preliminary studies suggest that alteration of the microbiome can help treat UC.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18-75 years of age.
* Established diagnosis of ulcerative colitis (UC) with known involvement of the left colon
* Mild to moderate disease defined as endoscopic evidence of disease with Mayo endoscopic sub-score 1 or 2 and total MAYO score ranging from 4-10. (The Mayo score ranges from 0 to 12, with higher scores indicating more severe disease. This score can be used for both initial evaluation and monitoring treatment response).
* Patients may be on any class of IBD-related medication (excluding steroids)
* Patients must be on stable medication regimen for at least 6 weeks prior to enrollment.
* Ability to understand and willingness to sign informed consent document

Exclusion Criteria:

* Patient who are asymptomatic
* Patients with severe, refractory disease (defined as Mayo scores of > 10, or endoscopic disease activity score of > 3) or patients with any other significant condition which, in the opinion of the investigator, could confound or interfere with evaluation of safety, tolerability of the investigational treatment or prevent compliance with the study protocol
* Prior colectomy
* Positive stool test for any of the following: Clostridium difficile by PCR, Salmonella, Shigella, Yersinia, Campylobacter, enteropathogenic E. coli by standard stool culture.
* Use of the steroid medications (any formulation) in the prior 6 weeks to enrollment
* Systemic antibiotic use within prior 6 weeks to enrollment
* Regular probiotic supplement use within prior 48 hours to enrollment
* Pregnancy or breastfeeding
* Severe immunodeficiency, inherited or acquired (e.g. HIV, chemotherapy, or radiation therapy)
* History of anaphylaxis (severe allergic reaction)
* Documented allergy to fluoroquinolones, metronidazole
* Life expectancy less than 12 months
* Age less than 18 or greater than 75 years of age
* History of esophageal or gastric motility disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Asses Endoscopic Stages of the Colon Pre/Post FMT | 2 years
  Assess endoscopic stage of the inflamed colon (endoscopic Mayo score) and assess the histologic stage of the biopsied colon (quiescent/mild/moderate/severe) pre and post FMT.
Asses Biologic Inflammatory Markers | 2 years
  Assess biologic inflammatory markers (ESR, CRP, fecal calprotectin, and fecal lactoferrin) pre and post FMT.
Review and Track Patient reported Outcomes via Validated Questionnaires | 2 Years
  Assess patient-report outcomes (symptomatology and quality of life) calculated via validated questionnaires (symptomatic Mayo Score and SF36)

SECONDARY OUTCOMES:
Change in metagenomic sequencing in Stool samples after FMT treatment | After 6, 12, and 18 Weeks
  Trace the effect FMT therapy has on microbiome diversity and to track whether this effect is sustained during and after therapy via metagenomic sequencing of stool samples at time 0, and weeks 6, 12, and 18.

OTHER OUTCOMES:
Asses changes in T-cell measures and serotonin signaling in mucosal biopsy samples and peripheral blood samples | 2 years
  Explore potential therapeutic mechanisms of FMT therapy. Changes in the host immune response before and after treatment will be assessed via measurement of both mucosal and peripheral T-cells populations (Th1, Th2, Th17) using mucosal biopsies and blood samples respectively.Changes in mucosal serotonin signaling will be measured using mucosal biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Moses, MD, Principal Investigator — The University of Vermont Medical Center
Locations (1):
- The University of Vermont Medical Center, Burlington, Vermont, United States

REFERENCES:
- [Derived] Crothers JW, Chu ND, Nguyen LTT, Phillips M, Collins C, Fortner K, Del Rio-Guerra R, Lavoie B, Callas P, Velez M, Cohn A, Elliott RJ, Wong WF, Vo E, Wilcox R, Smith M, Kassam Z, Budd R, Alm EJ, Mawe GM, Moses PL. Daily, oral FMT for long-term maintenance therapy in ulcerative colitis: results of a single-center, prospective, randomized pilot study. BMC Gastroenterol. 2021 Jul 8;21(1):281. doi: 10.1186/s12876-021-01856-9. PMID 34238227